CLINICAL TRIAL: NCT05148559
Title: Understanding and Addressing the Disparity in Vaccination Coverage Among U.S. Adolescents Living in Rural Versus Urban Areas
Brief Title: Impact of Adolescent Vaccine Reminder Notices Sent Via Preferred Method of Communication on HPV Vaccination
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huong Nguyen, PhD (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Huong Nguyen, PhD, Senior Research Scientist, Marshfield Clinic Research Foundation
Organization: Marshfield Clinic Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCL10517; U01IP001093 (NIH)
Record Dates: First submitted 2021-11-16; First posted 2021-12-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Reminder (Experimental)
  Interventions: Behavioral: Reminder Sent Via Preferred Method of Communication
- Standard of Care (Other)
  Interventions: Behavioral: Reminder Sent Via Mailed Letter

INTERVENTIONS:
Behavioral: Reminder Sent Via Preferred Method of Communication — Parents of 12 year-old patients due for ≥1 adolescent vaccine will receive a vaccine reminder notice every other month via their preferred method of communication (text message, email, mailed letter) until the adolescent receives all recommended vaccines, opts out of reminders, or turns 13.
  Arms: Enhanced Reminder
Behavioral: Reminder Sent Via Mailed Letter — Parents of 12 year-old patients due for ≥1 adolescent vaccine will receive a mailed vaccine reminder letter every other month until the adolescent receives all recommended vaccines, opts out of reminders, or turns 13.
  Arms: Standard of Care

SUMMARY:
Vaccine uptake in the United States is lower in rural areas, especially for HPV vaccine. Reminder/recall has been identified as an effective strategy to increase vaccination rates. This study will assess the impact by rurality of vaccine reminder notices sent via the parent's preferred method of communication on HPV vaccination among 12 year-old patients in a regional healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Marshfield Clinic Health System patient aged 12 years with at least one preventive visit or two evaluation & management visits with a Marshfield Clinic Health System provider in the last 36 months
* Due for at least one adolescent vaccine (HPV, MenACWY, Tdap)

Exclusion Criteria:

* Primary care provider is not affiliated with Marshfield Clinic Health System
* Opted out of Marshfield Clinic Health System vaccine reminder notifications
* Missing or invalid contact information
* Deceased

Ages: 12 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5451 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients that received 1 dose of HPV vaccine during follow-up based on electronic health data | 90 days
  Receipt of 1 dose of HPV vaccine within 90 days of receipt of reminder (yes/no) will be assessed using vaccination data available from the Marshfield Clinic Health System electronic health record, which includes vaccinations administered outside of MCHS through data exchanges with the Wisconsin Immunization Registry. Specifically patients will be classified as having received 1 dose of HPV vaccine if they have record of receipt of HPV vaccine with a vaccination date during the 90-day follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Huong McLean, PhD, Principal Investigator — Marshfield Clinic Research Institute
Locations (1):
- Marshfield Clinic Health System, Marshfield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT05148559/Prot_SAP_001.pdf